CLINICAL TRIAL: NCT00517478
Title: Thromboelastography As A Tool for Possible Clopidogrel Resistance in The Patients Treated With Primary PCI for STEMI
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Other Study IDs: 98/07
Record Dates: First submitted 2007-08-15; First posted 2007-08-17 (Estimated); Last update posted 2007-08-17 (Estimated); Status verified 2007-07

CONDITIONS: Myocardial Infarction; Cardiovascular Disease
MeSH Terms: conditions — Myocardial Infarction; Cardiovascular Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Blood Sample

SUMMARY:
Determine usefulness of thromboelastography (TEG) as a valuable tool in ex-vivo assessing platelet response to aspirin and clopidogrel (dual) treatment and on-treatment platelet reactivity during acute ST segment elevation myocardial infarction (STEMI) in an acute phase during primary PCI (PPCI) and also during recovery been on maintenance medical therapy and to determine the correlation between platelet response to clopidogrel treatment and the outcome of patients.

DETAILED DESCRIPTION:
Dual anti-aggregant therapy is recommended standard of therapy applicable to all patient groups undergoing PPCI. The aspirin-clopidogrel regiment is signed to every patient without assessing therapeutic effect. In face of growing evidence of platelet resistance to the standardized therapy there is a demand for reliable diagnostic tool for rapid and accurate assessment of platelet reactivity. TEG is an established technique to assess the quality of clot formation' used mainly in surgery and obstetrics to determine possible bleeding diathesis. Recently it became to be used in cardiology, where it can be a valuable tool to assess a response to antiplatelet therapy and its association with the outcome. However, there is a few data about use of TEG in STEMI patients undergoing PCI. Our study is designed to assess by TEG the platelet's response to clopidogrel treatment during acute STEMI in patients undergoing primary PCI and the correlation of this response with the long term outcome.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old STEMI patients admitted to ICCU and in whom the primary PCI is elected as treatment strategy would be enrolled

Exclusion Criteria:

* Patient received thrombolytic therapy, chronic renal failure (GFR<40 ml/min), any known hematological dyscrasia

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-08; Study Completion 2008-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Alex Blatt, MD, Study Director — Cardiology Division, Assaf Harofeh Medical Center; Ilia Litovchik, MD, Principal Investigator — Cardiology Division, Assaf Harofeh Medical Center
Locations (1):
- Asaf Harofeh MC, Ẕerifin, Zerifin, Israel